CLINICAL TRIAL: NCT07338149
Title: Detection of Syndesmotic Malreduction by Postoperative Computed Tomography in Ankle Fractures With Acceptable Radiographs: A Prospective Cohort Study
Brief Title: Postoperative Computed Tomography Detection of Syndesmotic Malreduction in Ankle Fractures
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Professor of Orthopedic Sugery, Cairo University
Other Study IDs: MS-310-2021
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Ankle Fractures
Keywords: Syndesmotic malreduction, Ankle fracture fixation, Computed tomography, Postoperative imaging, Functional outcome, AOFAS score
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ankle Fracture Patients With Syndesmotic Fixation: Adult patients with ankle fractures requiring operative fixation and syndesmotic stabilization who demonstrated acceptable postoperative plain radiographs and were followed prospectively for imaging and functional outcome assessment.

SUMMARY:
This prospective observational cohort study aims to evaluate the ability of postoperative plain radiographs to detect syndesmotic reduction accuracy in patients with ankle fractures requiring syndesmotic fixation. All included patients have acceptable postoperative radiographs according to standard radiographic criteria and undergo postoperative computed tomography to further assess syndesmotic reduction. Functional outcomes are assessed at one year following surgery using a standardized ankle functional score. The study seeks to explore the association between computed tomography-detected syndesmotic malreduction and postoperative functional outcome.

DETAILED DESCRIPTION:
Accurate reduction of the distal tibiofibular syndesmosis is essential for restoring ankle stability and achieving favorable functional outcomes after ankle fracture fixation. Plain radiographs are routinely used to assess postoperative syndesmotic reduction; however, subtle malreductions may not be detected using standard radiographic views alone.

This prospective observational cohort study includes adult patients with ankle fractures requiring operative fixation and syndesmotic stabilization who demonstrate acceptable postoperative plain radiographs. As part of postoperative evaluation, all included patients undergo computed tomography imaging to provide a more detailed assessment of syndesmotic reduction, particularly with respect to rotational and translational alignment of the distal fibula relative to the tibia.

Based on computed tomography findings, syndesmotic reduction is categorized according to predefined criteria. Functional outcomes are assessed at 12 months postoperatively using the American Orthopaedic Foot and Ankle Society ankle-hindfoot score. The study is observational in nature, and imaging findings do not influence postoperative management or treatment decisions.

The objective of this study is to assess the limitations of plain radiographs in detecting syndesmotic malreduction and to evaluate the association between computed tomography findings and functional outcomes following ankle fracture fixation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Acute ankle fractures requiring operative fixation with syndesmotic stabilization
* Acceptable postoperative plain radiographs based on standard radiographic criteria
* Ability to comply with follow-up and functional assessment

Exclusion Criteria:

* Open ankle fractures
* Previous surgery on the affected ankle
* Polytrauma patients
* Pathological fractures
* Incomplete imaging or follow-up data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute ankle fractures requiring operative fixation and syndesmotic stabilization who demonstrated acceptable postoperative plain radiographs and were prospectively followed for postoperative imaging assessment and functional outcome evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Functional outcome assessed by the American Orthopaedic Foot and Ankle Society ankle-hindfoot score | 12 months postoperatively
  Functional outcome of the affected ankle assessed using the American Orthopaedic Foot and Ankle Society (AOFAS) ankle-hindfoot score, which evaluates pain, function, and alignment on a 0-100 point scale, with higher scores indicating better function.

SECONDARY OUTCOMES:
Syndesmotic reduction accuracy assessed by postoperative computed tomography | within 1 week after surgery
  Accuracy of distal tibiofibular syndesmotic reduction assessed using postoperative computed tomography imaging, based on predefined radiological criteria evaluating translational and rotational alignment of the distal fibula relative to the tibia.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No